CLINICAL TRIAL: NCT07257848
Title: Practice-Based Evidence in Ecuador: Routine Monitoring of Outcomes and Change in Psychotherapy for Common Mental Health Problems
Brief Title: Practice-Based Evidence in Psychotherapy: A Multicentric Study From Ecuador
Acronym: CLIP_Ecuador
Status: Recruiting | Type: Observational
Sponsor: Universidad de las Americas - Quito (Other)
Responsible Party: Principal Investigator, Clara Paz, Researcher, Universidad de las Americas - Quito
Other Study IDs: 2024-OBS-033
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Psychological Distress
Keywords: practice-based evidence; routine outcome monitoring; psychotherapy; practice-oriented research; change; outcome; psychological distress; Latin America; Practice Research Network; Consorcio Latinoamericano de Investigación en Psicoterapia
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Helpseeking Ecuadorian adult and adolescent clients: The participants will consist of adolescent (ages 11-17) and adult (ages 18 and above) clients who present with common, non-severe mental health problems and are seeking services at the participating clinics involved in this study.
  Interventions: Behavioral: Psychological Intervention

INTERVENTIONS:
Behavioral: Psychological Intervention — Real-world application of psychological care, adapted to the individual needs of clients within the normal workflow of clinical practice. Treatments are delivered by licensed practitioners in routine clinical settings, ensuring that interventions are tailored to each client's specific characteristics and therapeutic goals.

SUMMARY:
The goal of this observational study is to learn about the progress and outcomes of clients receiving psychotherapy for common mental health problems in Ecuador. The main questions it aims to answer are:

* How much do clients' psychological distress typically change during the course of their psychotherapy?
* What factors are associated with outcomes in real-world mental health services in Ecuador?

This study involves clients who are about to start psychotherapy at one of the participating mental health clinics in Ecuador. Participants will continue their regular psychotherapy sessions as usual. The only addition is that before their sessions, they will be asked to complete questionnaires about their general well-being. This routine check-in process will continue throughout their time in therapy. Contextual information will be collected before starting treatment, and satisfaction with the treatment and any contextual changes will be collected after treatment ends.

DETAILED DESCRIPTION:
This project is an exploratory, descriptive, and longitudinal naturalistic study. Its primary objective is to systematically examine client progress and treatment outcomes across a network of psychological care services in Ecuador by implementing a Routine Outcome Monitoring system. As a naturalistic investigation, the study will be conducted within existing clinical settings, ensuring that findings reflect real-world therapeutic practices with adolescent and adult populations.

The research will be implemented across multiple psychological care centers throughout Ecuador. To provide a comprehensive understanding of therapeutic processes, data will be collected at three distinct levels. At the client level, psychological distress serves as the primary outcome variable, supplemented by sociodemographic information collected at pre-treatment and post-treatment intervals and treatment satisfaction measures at post-treatment. At the therapist level, clinicians will complete client intake forms at treatment initiation and personal style questionnaires at treatment conclusion. Additionally, service-level data will be gathered from each participating center to characterize operational contexts and organizational frameworks.

The anticipated outcomes of this initiative are substantial. It will establish systematic tracking of client progress throughout therapy, enabling identification of population-specific levels of psychological distress and change trajectories. Furthermore, the project aims to create a foundational framework for the widespread implementation of outcome measurement systems in Ecuador's mental health care context.

In the long term, this project seeks to promote the consistent and generalized adoption of Routine Outcome Monitoring systems, thereby contributing to the development of a Practice-Based Evidence culture in Ecuador and throughout Latin America. It will strengthen Practice-Based Research Networks in psychological interventions, particularly through collaboration with established organizations such as the Consorcio Latinoamericano de Investigación en Psicoterapia (CLIP), fostering regional cooperation and standardizing assessment methodologies across mental health services.

ELIGIBILITY:
Clients

Inclusion Criteria:

* Be 11 years of age or older.
* Have sufficient ability to communicate in Spanish.
* Undergo psychological treatment at one of the mental health services included in the project.

Exclusion Criteria:

* Present substantial cognitive deficits that do not allow the development of the evaluation.

Therapists

Inclusion Criteria:

* Therapist providing psychological treatment at one of the mental health services included in the project.

Supervisors

Inclusion Criteria:

* Provide clinical supervision to therapists delivering treatment at any of the project's affiliated mental health services.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participant pool will consist of three groups: (1) help-seeking clients engaged in treatment, (2) therapists providing services, and (3) supervisors from the project's affiliated mental health services in Ecuador.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) | At baseline and immediately after treatment completion
  The CORE-OM is a 34-item self-report instrument designed for use across heterogeneous services and grounded in a pan-theoretic core of psychological distress, including subjective well-being, problems, risk, and functioning. Items are scored on a scale from 0 (never) to 4 (always or almost always). Higher scores indicate greater psychological distress. This instrument is suitable as an initial assessment tool and as an outcome measure. The Spanish version of this measure will be used. This version was translated in Spain and has shown good psychometric properties in Spain and Ecuador. CORE-OM is administered to adult clients.
Change in Clinical Outcomes in Routine Evaluation-10 (CORE-10) | From the second treatment session through treatment completion (an average of 10 weeks)
  The CORE-10 is a generic, short, and easy-to-use assessment measure. Its items were drawn from the CORE-OM. The CORE-10 is an instrument that has shown good psychometric properties and is practical for use on a session-by-session basis with people presenting with psychological distress in mental health settings. Its Spanish version will be used. In Ecuador, this version has shown good psychometric properties. CORE-10 is administered to adult clients.
Change in Young Person's-Clinical Outcomes in Routine Evaluation (YP-CORE) | From baseline through treatment completion (an average of 10 weeks)
  The YP-CORE is a brief self-report instrument capable of detecting psychological distress in adolescents, generated by a wide range of problems, while providing information about the person's general functioning. It has 10 items, which must be answered on a 5-point scale (0 to 4). Its Spanish version will be used. The YP-CORE was translated into Spanish and showed adequate psychometric properties. In the present study, we will use a version of this measure, adapted for Ecuador and Latin America, which has good psychometric properties in Ecuador. YP-CORE is administered to adolescents.

SECONDARY OUTCOMES:
Emotional and Psychological Outcome (EPO-1) | From Baseline through treatment completion (an average of 10 weeks)
  The EPO-1 is a single-item outcome measure in which clients assess their current emotional and psychological state by responding to the question: "At this moment, how are you doing emotionally and psychologically?" This item is scored on a 5-point scale ranging from 0 ("Very bad; I can barely handle things") to 4 ("Very well; I have no significant complaints"). EPO-1 is administered to all clients.
Satisfaction with the Treatment Received Scale (CRES-4) | At the treatment completion visit, approximately 10 weeks post-enrollment.
  The CRES-4 scale has 4 items: one question on satisfaction, one on the level of resolution of the main problem, one on emotional state before the start of treatment, and one on emotional state when completing the questionnaire. These questions allow interpretations of the perceived change in their emotional state, satisfaction, and problem resolution. In this study, the Spanish version of this measure will be used.CRES-4 is administered to all clients.

OTHER OUTCOMES:
CORE Therapy Assessment Form (CORE-A-TAF) | CORE-A-TAF is completed by the therapists at baseline
  The CORE-A-TAF is a pragmatic form intended to be completed by therapists at baseline. The CORE-TAF includes referral information, sociodemographic data on the client, and data on the nature, severity, and duration of the client's problems. We will use its Spanish version, which is currently being translated and adapted for use by the CLIP.
CORE End of Therapy (CORE-A-EoT) | CORE EoT is completed by the therapists immediately after treatment completion
  The CORE-A-EoT is a pragmatic form designed to be filled out by therapists immediately after treatment completion. The CORE-A-EoT reports on the completed treatment, including the number of sessions, type of therapy, length and frequency of sessions, whether the ending was planned or unplanned, and the potential benefits of therapy. We will use its Spanish version, which is currently being translated and adapted for use by the CLIP.
Assessment questionnaire on the personal style of the therapist (PST-Q) | Baseline (Enrollment), 12 months, 24 months, and 36 months.
  The PST-Q is a 20-item self-report instrument with a 7-point Likert scale (1 "Completely Disagree" to 7 "Completely Agree"). It assesses the therapist's position across five dimensions: instructional, expressive, involvement, attentional, and operative. Therapists will complete the PST-Q.
Service Information Form | Baseline (Enrollment), 12 months, 24 months, and 36 months.
  This form is intended to be completed by the supervisors or authorities of each service. It collects general data about the center, such as the type of population it serves, its annual average number of users, etc. Supervisors will complete this form.

CONTACTS AND LOCATIONS:
Locations (11):
- Ecuador (11):
  - Centro de Psicología Aplicada, Universidad de Las Américas, Ecuador, Quito, (P)Pichincha
  - Jorge López Consultorios, Manta, Manabí
  - PsicoNeuro Manta, Manta, Manabí
  - Historie, Quito, Pichincha
  - Kumpana, Quito, Pichincha
  - Mentis Psicología, Quito, Pichincha
  - Equimente, Quito, Pichincha
  - Sentir Psicología Integral, Quito, Pichincha
  - Solo Psique, Quito, Pichincha
  - Renova - Mentis Habitus Positive, Quito, Pichincha
  - Psico Estratégico, Quito, Pichincha

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valdiviezo-Ona J, Ortiz-Mancheno N, Valdivieso-Arias G, Erazo-Perez D, Rodriguez-Lorenzana A, Evans C, Paz C. Assessing the suitability and psychometric properties of the Spanish version of the YP-CORE for adolescents in Latin America: a study in Ecuador. BMC Psychol. 2024 Nov 18;12(1):671. doi: 10.1186/s40359-024-02169-8. PMID 39558391
- [Background] Paz C, Mascialino G, Proano K, Evans C. Psychological intervention change measurement in Latin America: Where from? Where to? Psychother Res. 2021 Jan;31(1):132-141. doi: 10.1080/10503307.2020.1750728. Epub 2020 Apr 16. PMID 32297845
- [Background] Trujillo A, Feixas G, Bados A, Garcia-Grau E, Salla M, Medina JC, Montesano A, Soriano J, Medeiros-Ferreira L, Canete J, Corbella S, Grau A, Lana F, Evans C. Psychometric properties of the Spanish version of the Clinical Outcomes in Routine Evaluation - Outcome Measure. Neuropsychiatr Dis Treat. 2016 Jun 21;12:1457-66. doi: 10.2147/NDT.S103079. eCollection 2016. PMID 27382288
- [Background] Paz C, Mascialino G, Evans C. Exploration of the psychometric properties of the Clinical Outcomes in Routine Evaluation-Outcome Measure in Ecuador. BMC Psychol. 2020 Sep 1;8(1):94. doi: 10.1186/s40359-020-00443-z. PMID 32873334
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Valdiviezo-Ona J, Montesano A, Evans C, Paz C. Fostering practice-based evidence through routine outcome monitoring in a university psychotherapy service for common mental health problems: a protocol for a naturalistic, observational study. BMJ Open. 2023 May 24;13(5):e071875. doi: 10.1136/bmjopen-2023-071875. PMID 37225267
- See also: MarBar is the system used for data collection in all the mental health services involved in the study — https://www.marbarsystem.com/
- See also: Clinical Outcomes in Routine Evaluation meeasures information — https://www.coresystemtrust.org.uk/